CLINICAL TRIAL: NCT06800885
Title: Repeated Cross Sectional Surveillance Study To Determine the Influenza Vaccination Rates in German Participants During Current Respiratory Season
Brief Title: Repeated Cross Sectional Surveillance Study To Determine the Influenza Vaccination Rates in German Participants
Acronym: Vakzimeter FLU
Status: Active, not recruiting | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: FLU00216
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Influenza Immunization
Keywords: Seasonal Influenza; Influenza Vaccination Rates
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: 18 Years of Age to 59 Years of age: Healthy diverse adults aged 18 years to 59 (inclusive) years of age
- Group 2: 60 Years of Age and Older: Healthy diverse adults aged 60 years (inclusive) of age and older
- Subgroup 1: Pregnant Women 18 Years of Age to 59 Years of Age: Pregnant woman aged 18 years to 59 (inclusive) years of age
- Subgroup 2: Patients with Chronic Illness: Diverse patients with chronic illness

SUMMARY:
Real-time monitoring of vaccination rates for Germany is unavailable, and up-to-date data publication is delayed, which makes it challenging to develop effective public health strategies to increase vaccination coverage.

This study aims to address the gap by assessing current influenza vaccination rates, particularly among those aged 60 and older, to inform public health interventions and encourage healthcare providers to recommend influenza vaccination more proactively.

The primary objective of this study is to determine the influenza vaccination rates in the German population during the current respiratory season. The study will focus on:

1. Assessing the vaccination rates among the two main age groups 18 years of age through and including 59 years of age and 60 years of age (inclusive) and older
2. Assessing the vaccination rate among individuals with risk-based vaccination recommendation according to Standing Committee on Vaccination (Ständige Impfkommission) (STIKO) The study will target a disproportionate sample of the German population regarding age: 30% aged 18 years of age through and including 59 year of age and 70% aged 60 years of age (inclusive) and older. Within these age groups, the study targets a representative distribution regarding gender and region.

This study is conducted as an online survey that will either be self-completed by the respondents (CAWI) or completed via an interviewer for a subgroup of respondents aged 70+ (CATI). The survey is estimated to last 10 minutes and will comprise of closed-ended questions only (i.e., respondents will not have the possibility to add any free-text). The survey will be conducted in German.

The panelists will be divided into strata based on demographic variables like gender and region. Within each stratum, participants will be randomly selected to participate in the survey.

ELIGIBILITY:
Inclusion Criteria:

* Reside in Germany at the time of survey completion
* Be at least 18 years old at the time of survey completion.
* Agree with privacy policy and AE (Adverse Event) reporting requirements before proceeding with the survey.
* Read and agree to the ICF (Informed Consent Form) by ticking a box before proceeding with the survey or telephone interview.

Exclusion Criteria:

* Participation in the study (= completed the survey or telephone interview) in a previous wave of the current season.
* Living in nursing home Note: The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The number of participants surveyed will be approximately 6,000 per season using CAWI. These are spread over a total of 6 waves per season, resulting in a sample size of 1,000 respondents per wave using CAWI.
  The study will target a disproportionate sample of the German population regarding age: 30% aged 18 years of age though and including 59 years of age and 70% aged 60 years of age and older. Within these age groups, the study targets a representative distribution regarding gender and region.
  This study is conducted as an online survey that will either be self-completed by the respondents (CAWI) or completed via an interviewer for a subgroup of respondents aged 70+ (CATI). The survey is estimated to last 10 minutes and will comprise of closed-ended questions only (i.e., respondents will not have the possibility to add any free-text). The survey will be conducted in German.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Assessing the seasonal influenza vaccination rates among diverse healthy participants 18 years of age through and including 59 years of age | Throughout Study (Approximately 3 months)
  Descriptive analysis of vaccination status (yes/no) will be performed using summary statistics, i.e., proportion of vaccinated individuals among all enrolled persons per wave in the age group 18 years of age to and including 59 years of age
Assessing the seasonal influenza vaccination rates among diverse healthy participants 18 years through and including 34 years of age | Throughout Study (Approximately 3 months)
  Descriptive analysis of vaccination status (yes/no) will be performed using summary statistics, i.e., proportion of vaccinated individuals among all enrolled persons per wave in the age group 18 years of age through 34 years of age
Assessing the seasonal influenza vaccination rates among pregnant women (with or without co-morbidities) | Throughout Study (Approximately 3 months)
  Descriptive analysis of vaccination status (yes/no) will be performed using summary statistics, i.e., proportion of vaccinated individuals among all enrolled persons per wave in pregnant women with or without co-morbidities
Assessing the seasonal influenza vaccination rates among diverse patients with chronic illness | Throughout Study (Approximately 3 months)
  Descriptive analysis of vaccination status (yes/no) will be performed using summary statistics, i.e., proportion of vaccinated individuals among all enrolled persons per wave in diverse patients with chronic illness
Assessing the seasonal influenza vaccination rates among diverse healthy participants 35 years through and including 59 years of age | Throughout Study (Approximately 3 months)
  Descriptive analysis of vaccination status (yes/no) will be performed using summary statistics, i.e., proportion of vaccinated individuals among all enrolled persons per wave in the age group 35 years of age through and including 59 years of age
Assessing the seasonal influenza vaccination rates among diverse healthy participants 18 years through and including 59 years of age | Throughout Study (Approximately 3 months)
  Descriptive analysis of vaccination status (yes/no) will be performed using summary statistics, i.e., proportion of vaccinated individuals among all enrolled persons per wave in the age group 18 years of age through and including 59 years of age
Assessing the seasonal influenza vaccination rates among diverse healthy participants older than 60 years of age | Throughout Study (Approximately 3 months)
  Descriptive analysis of vaccination status (yes/no) will be performed using summary statistics, i.e., proportion of vaccinated individuals among all enrolled persons per wave in the older than 60 years of age group
Assessing the seasonal influenza vaccination rates among diverse healthy participants aged 60 years of age through and including 69 years of age | Throughout Study (Approximately 3 months)
  Descriptive analysis of vaccination status (yes/no) will be performed using summary statistics, i.e., proportion of vaccinated individuals among all enrolled persons per wave in the age group 60 years of age through and including 69 years of age
Assessing the seasonal influenza vaccination rates among diverse healthy participants aged 70 years of age through and including 79 years of age | Throughout Study (Approximately 3 months)
  Descriptive analysis of vaccination status (yes/no) will be performed using summary statistics, i.e., proportion of vaccinated individuals among all enrolled persons per wave in the age group 70 years of age through and including 79 years of age
Assessing the seasonal influenza vaccination rates among diverse healthy participants older than 80 years of age | Throughout Study (Approximately 3 months)
  Descriptive analysis of vaccination status (yes/no) will be performed using summary statistics, i.e., proportion of vaccinated individuals among all enrolled persons per wave in the older than 80 years of age group

SECONDARY OUTCOMES:
Assessing the seasonal evolution of the influenza vaccination coverage rates (VCR) among the two main age groups 18 years of age through and including 59 years of age and 60 years of age and older (inclusive) | Throughout Study (approxmatley 3 months)
  Descriptive analysis of VCR by time of survey during the season (as proportion of vaccinated individuals among all enrolled persons per wave in the two main age groups 18 year of age through and including 59 years of age and 60 years of age (inclusive) and older, and per subgroup/strata)
Assessing the seasonal evolution of the influenza vaccination coverage rates (VCR) through time trends among the two main age groups 18 years of age through and including 59 years of age and 60 years of age and older (inclusive) | Throughout Study (approxmatley 3 months)
  Analysis of time trends over the three seasons, based on VCR data collected in January of each year (last wave) (as proportion of vaccinated individuals among all enrolled persons per wave in the two main age groups 18 year of age through and including 59 years of age and 60 years of age (inclusive) and older, and per subgroup/strata)
Assessing reasons for/against influenza vaccination in the target population of the STIKO recommendation for each season | Throughout study (approximatley 3 months)
  Descriptive analysis of vaccination status (yes/no) and reasons for or against influenza vaccination will be performed using summary statistics, i.e., proportion of vaccinated individuals among all enrolled persons per wave in the two main age groups 18 year of age through and including 59 years of age and 60 years of age (inclusive) and older, and per subgroup/strata)
Assess the reliability of a demographic study based on randomly sampled population groups using Computer-Assisted Web Interview (CAWI) for estimating VCR | Throughout the study (approximatley 3 months)
  Descriptive analysis of VCR (proportions) for the two main age groups 18 years of age through 59 and 60 years (inclusive) of age and older and per subgroup/strata) in comparison with results from the Robert Koch-Institute (RKI) vaccination surveillance
Compare the reliability of VCR estimates in the elderly population (70+ years) obtained through a mixed approach of CAWI and Computer assisted telephone interview (CATI) versus CAWI only (in the first season) | Throughout the study (approximatley 3 months)
  Descriptive analysis of VCR (proportions) in the regions with mixed mode data collection approach in comparison with other regions and with results from the RKI vaccination surveillance for age group 70 years of age and older

CONTACTS AND LOCATIONS:
Locations (1):
- Germany, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org